CLINICAL TRIAL: NCT03256682
Title: The Efficacy of a Mobile Video Counseling Targeted for Stress Reduction and Resilience Enhancement in Employees With Emotional Labor
Brief Title: The Efficacy of Mobile Video Counseling for Employees With Emotional Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Trade, Industry & Energy, Republic of Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-1707-408-305
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2017-07

CONDITIONS: Stress, Psychological
Keywords: Resilience; Mobile video counseling; Emotiona labor
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Healthy individuals recruited through advertisement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobile Video Counseling (Experimental): Utilize mobile imaging equipment, receive a total of 4 stress management consultations every 50 minutes at a time, once a week.
  Interventions: Behavioral: Stress management counseling
- Offline Counseling (Active Comparator): Receive a total of 4 stress management counseling, once a week for 50 minutes each session.
  Interventions: Behavioral: Stress management counseling
- Selfcare (No Intervention): Use stress management materials to manage yourself.

INTERVENTIONS:
Behavioral: Stress management counseling — stress management counseling based on CBT and relaxation
  Arms: Mobile Video Counseling; Offline Counseling

SUMMARY:
The purpose of this study is to verify the effectiveness of mobile video counseling for workers. Subjects who can participate in the screening evaluation are assigned to one of face-to-face counseling group, mobile counseling group, and self-treatment group. The mobile counseling group and the face-to-face counseling group counseld with a total of 4 times, 50 minutes at a time, once a week, and the self-treatment group provides self-education by providing the stress education kit.

DETAILED DESCRIPTION:
After screening, Pre-evaluation is conducted on the subjects who agreed to participate in the study. Pre-assessment includes questionnaires related to stress, emotional labor, resilience, sleep, etc., and includes stress-related physiological measures using HRV, 2 lead EEG. After the pre-evaluation, the test group will conduct a counseling program with a psychologist for 50 minutes at a time, once a week, for a total of 4 sessions (one month for a period). The place should be placed in a quiet place where the subject thinks comfortably and is designated as the same place to exclude the influence by the place, but the subject does not have to visit the hospital. In the offline counseling group, four counseling sessions are held with the psychologist off-line for a total of 4 counseling sessions, 50 minutes at a time, once a week after the same pre-evaluation. As a self-care control, counseling is not provided and self-learning materials are provided once a week.

Mobile counseling group and offline counseling group visit the hospital within one week after termination and within 4 to 5 weeks after pre-evaluation in self-care control group. Also, to see if the effect of mobile counseling is continued even after counseling is completed, visit the counseling clinic one month after counseling is over and conduct the same test. The data obtained from this study showed that the mobile counseling program measured the change in the clinical scale and heart rate variability and EEG such as the stress and resilience of the subjects, and the self-care group using the offline counseling group and stress data and stress related psychological and physiological And compare the effects on the improvement of the indicator.

ELIGIBILITY:
Inclusion Criteria:

* Workers over the age of 19 and under 65
* In the Perceived Stress Scale 14 points or more
* If you are currently taking medication due to psychiatric illnesses such as depression, anxiety disorder, insomnia, etc., if the stabilizer is expected to have no change in drug dose during the clinical trial
* If you understand the protocol and voluntarily agree to participate
* If you have an Android phone

Exclusion Criteria:

* Age under 19, adult over 65
* If you have dementia, intellectual disability, or other cognitive impairment
* If you have convulsive disorder, stroke, or other neurological disorder
* If you have psychosis such as schizophrenia or bipolar disorder or you have a history
* If you have a disease that can affect the reliability of HRV test, such as heart disease or lung disease.
* Has received non-pharmacological psychiatric or counseling treatment within the current or last 6 months.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline Perceived Stress Scale (PSS) score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  14-item scale developed by Cohen et al. (1983) that emphasizes subjective perception of stress. Measures the degree of perceived unforeseeable, uncontrollable, and overwhelming experience of stress in the past month.

SECONDARY OUTCOMES:
Change from baseline Korean Emotional Labor Assessment Tool score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  The total of 26 items were Emotional expression and control 5 items, organizational monitoring and management system 4 items, forced customer response 4 items, emotional damage 6 items, organizational protection system 7 items, and organizational protection system is reverse coding and summed up. 4 point Likert scale (1 = not at all, 5 = very much), and the possible total score ranges from 26 to 130 points. The higher the score, the more emotional labor means.
Change from baseline Korean abbreviation of Occupational Stress Scale (KOSS) score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  total of 24 items were used, and each item was not at all (from 1 point) to very much (5 points). The higher the score, the more the job stress means. Job demand, Insufficient job control, job insecurity, interpersonal conflict, Organizational system, Lack of reward and Occupational climate.
Change from baseline Patient Health Questionnaire 9 (PHQ-9) score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  The total score is 0 to 27, and the higher the total score, the more severe the depressive symptoms. Cutpoints of 5, 10, 15 and 20 represent the thresholds for mild, moderate, moderate severe, and severe depression, respectively.
Change from baseline Brief resilience scale (BRS) score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  It is composed of 6 questions and is evaluated on the 5-point scale (1: not at all, 5: very much)
Change from baseline Athens Insomnia Scale (AIS) score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  total score of 6 points was used as a breakpoint, this Using the quality index of Pittsburgh Sleep, which is widely used to evaluate the quality of sleep
Change from baseline Depression, Anxiety, Stress Scale (DASS) score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  A total of 21 questions, depression, anxiety, and stress were assessed on a 4-point scale (0: not at all, 3: very or almost always). In this study, only 7 items relating to anxiety were extracted. The lowest score is from 0 to the maximum score of 21, and the higher the score, the more severe anxiety. Anxiety scores above 8 indicate significant anxiety symptoms
Change from baseline Connor-Davidson Resilience Scale (CD-RISC) score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  A total of 25 items were assessed as a 5-point Likert scale (0: not at all, 4: very much). A score of 0-100 means higher resilience
Change from baseline Maslach Burnout Inventory-General Survey (MBI-GS) score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  Evaluate on a total of 16 questions on a 7 point scale (1 point = not at all, 7 points = very much). The higher the total score, the greater the degree of job exhaustion.
Change from baseline Heart rate variability (HRV) and Change from baseline Eletroencephalogram (EEG) score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  The instrument measures the EEG from the headset forehead sensor (EEG measurement of the prefrontal lobe, 2 channel EEG) and measures the pulse at the earlobe (measure the pulse rate in the earlobe vessel using a light sensor). The results of EEG and heart rate variability were calculated by measuring for 5 minutes.

OTHER OUTCOMES:
Counseling Satisfaction Scale | After 4 weeks intervention
  Evaluate within 7 days of closing psychological counseling. Twelve questions to evaluate the quality of psychological counseling, content, psychological counselor 's attitude, procedures, and six questions to measure accessibility and a written description question for the proposal. The mobile group further includes questions such as system speed, image quality, sound and so on. Evaluating from not at all (1 point) very much (5 points), which means that the higher the score is, the higher the degree of satisfaction is.
Change from baseline Working Memory score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  Measure short-term memory, work function known to be sensitive to stress. It consists of forward, backward, sequencing, scored 0 - 14 points, and means that the higher the score, the better the function.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hyun Kim, MD, Ph.D, Principal Investigator — Seoul National Univerysity Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860
- [Derived] Kim JI, Yun JY, Park H, Park SY, Ahn Y, Lee H, Kim TK, Yoon S, Lee YJ, Oh S, Denninger JW, Kim BN, Kim JH. A Mobile Videoconference-Based Intervention on Stress Reduction and Resilience Enhancement in Employees: Randomized Controlled Trial. J Med Internet Res. 2018 Oct 22;20(10):e10760. doi: 10.2196/10760. PMID 30348630